CLINICAL TRIAL: NCT03698760
Title: Calibration and Validation of a Computerized Olfactory Test in Subjects With Alzheimer's Disease in a Mild Stage
Brief Title: Computerized Olfactory Test - Alzheimer Disease Mild Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1509
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease; Olfaction Disorders
MeSH Terms: conditions — Alzheimer Disease; Olfaction Disorders

STUDY DESIGN:
Intervention Model Description: The study is a single-center controlled study (Jewish General Hospital, Montreal, Quebec, Canada), consisting of two groups of subjects: a control group and a group of subjects with mild Alzheimer's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild stage Alzheimer group (Experimental): Participants with mild stage Alzheimer's disease
  Interventions: Diagnostic Test: Olfactory test
- Control Group (Experimental): Participants without cognitive disorders
  Interventions: Diagnostic Test: Olfactory test

INTERVENTIONS:
Diagnostic Test: Olfactory test — Olfactory test:
  All fragrances tested are kept in an airtight case protected from cold and heat.
  The test is done on a tablet and the data will be automatically saved. The first screen is about the administrative data, sex and age of the subject. Olfactory test: six odors among the fourteen are proposed in a randomized way.

SUMMARY:
This study evaluates the effectiveness of the smell tests that are used in early diagnosis of mild dementia.

DETAILED DESCRIPTION:
For twenty years research has shown a strong link between olfactory disorders and Alzheimer's disease. The focus is on the very early alteration of the olfaction which acts as a harbinger of the disease since it is detectable in its asymptomatic phase. In addition, olfactory involvement is a precursor to the transformation of mild cognitive impairment into MA. Indeed the anatomical structures the first lesions are located in the transentorhinal region of the temporal lobe and entorhinal phase, before progressing towards the limbic system, which will mark the clinical appearance of the first signs of AD.

In literature, it has been shown that there was no olfactory test that is recognized as a gold standard in the scientific community due to a lack of homogeneity of the tools used, their availability and their validity depending on the culture. Moreover, of all the tests currently available, none are specific to neurodegenerative diseases.

Very recent studies show that there is also a strong preference for imaging tools or biomarkers in the detection of AD, but it appears that the olfactory disorders are well before these markers. It has been shown that an identification test is comparable in predictive accuracy to neuroimaging and cerebrospinal fluid sampling.

This study will therefore focus on the calibration and validation of a computerized olfactory test for the diagnosis of Alzheimer's disease and based the recommendations of professionals so as to promote the effective use of this test in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years old and over
* The participants enrolled in the control group must have a score of the Mini-Mental State Exam test greater than or equal to 28.
* The participants enrolled in the intervention group must have a diagnosis of Alzheimer's disease, and the score of the Mini-Mental State Exam test should be between 20 and 27

Exclusion Criteria:

* Presenting an unstable, acute or current psychiatric or physical condition that is severe enough to prevent the participant from participating in the study, as determined by the investigator.
* Having an uncorrected major visual or hearing impairment or anosmia (total olfaction loss).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Objective test of evaluation of the olfactory sensitivity | 15 minutes
  olfactory test (only one evaluation): random fragrances, recognition (Yes or No)

SECONDARY OUTCOMES:
Health condition assessed by self-administered questionnaire (SAQ) | 10 minutes
  self-administered questionnaire (SAQ), score between 0 and 18, a higher score means a higher frailty
Objective test of evaluation of the olfactory thresholds | 15 minutes
  olfactory test, 6 random fragrances among 14, recognition Yes or No and at what concentration

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada